CLINICAL TRIAL: NCT03502317
Title: Prehabilitation to Improve Cancer Surgery Outcomes (PICaSO): A Randomized Controlled Trial
Brief Title: Prehabilitation to Improve Cancer Surgery Outcomes
Acronym: PICaSO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-0185
Record Dates: First submitted 2018-03-25; First posted 2018-04-18 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Gastrointestinal Cancer; Prehabilitation; Surgery; Physical Activity
Keywords: Prehabilitation; Gastrointestinal Cancer; Physical Activity; Exercise; Surgery
MeSH Terms: conditions — Gastrointestinal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Study Arm (Experimental): Patients will participate in a two-pronged prehabilitation strategy - physical prehabilitation and psychological prehabilitation. Prehabilitation will last from a minimum of 21 days to a maximum of 42 days before a patient's clinically indicated surgery.
  Interventions: Behavioral: Physical Prehabilitation; Behavioral: Psychological Prehabilitation
- Usual Care Study Arm (No Intervention): No specific exercises or stress reduction techniques are prescribed and the patient will be counseled to continue their current level of activity, and will be given the information on exercise as outlined in the Cancer Care Ontario guidelines. Patients in the Usual Care arm will also be given the same Fitbit activity tracker as patients in the Prehabilitation arm in order to eliminate the activity tracker as an intervention itself and to be able to track the activity (steps) for comparison. Patients in the Usual Care arm will be required to wear their Fitbit activity tracker from the day of randomization to 90 days post-surgery. Patients will record their steps in the diary provided.

INTERVENTIONS:
Behavioral: Physical Prehabilitation — Physical prehabilitation will comprise a personalized, home-based exercise program designed to meet the Cancer Care Ontario Exercise Guidelines for Cancer Survivors. A Registered Kinesiologist (RKin) will complete a baseline physical assessment and prescribe an individualized multi-modal exercise program consisting of 4-5 days of 30+ minutes of aerobic exercise (brisk walking or equivalent to target heart rate of 40-60% of max) and 2-3 days of moderate intensity resistance training of major muscle groups (8-10 repetitions). Participants will be provided with a Fitbit with a heart rate monitor, resistance bands, and a stability ball. Patients will be required to wear their Fitbit and record the number of steps at the end of each day from randomization to 90 days post-surgery.
  Arms: Prehabilitation Study Arm
Behavioral: Psychological Prehabilitation — Psychological prehabilitation will consist of one in-person coaching session of a 'mindfulness' informed intervention conducted by a specially trained RKin. The 40 minute coaching session will include a guided mindfulness session and debriefing. Participants will be asked to practice for 20 minutes twice a day. The patients will be given access to an audio file that will walk them through the 20 minute sessions.
  Arms: Prehabilitation Study Arm

SUMMARY:
This is a randomized control trial aiming to investigate the use of a prehabilitation regimen for patients undergoing major GI cancer surgery and its effects on measurements of HRQOL, LOS, and post-operative complications. Participants will be randomized to either the Prehabilitation arm or the Usual Care arm (control group). The Prehabilitation arm will be prescribed both physical and psychological prehabilitation prior to undergoing surgery for their GI cancer. The Usual Care arm will be counseled to continue their current level of activity and given the information on exercise as outlined in the Cancer Care Ontario guidelines. Participants in the Usual Care arm will also be given the same activity tracker as patients in the Prehabilitation arm in order to eliminate the activity tracker as an intervention itself. Clinical, patient-reported outcomes and health system outcomes will be evaluated. Outcomes will be measured at consent (baseline), immediately preoperatively, and postoperatively at 1, 3 and 6 months. The investigators will collect measures of recruitment, attrition and self-reported compliance via a log completed by the coordinator during weekly patient phone calls.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Fluent in English
* Able to comply with study procedures & follow-up contained within the consent form
* Pathologically or radiologically confirmed diagnosis of a GI cancer
* GI cancer must be considered operable
* Expected LOS ≥ 5 days as calculated by the validated American College of Surgeons Surgical Risk Calculator
* > 21 days between time of randomization and time of expected surgery
* Patient written, informed consent obtained according to ICH GCP guidelines and local regulations

Exclusion Criteria:

* < 18 years old
* Not fluent in English
* Planned resection of bony pelvis, limbs, or major lower extremity neurovascular structures
* Significant comorbidity including any of the following:

  * Canadian Cardiovascular Society class III/IV coronary disease
  * New York Heart Association class III/IV congestive heart failure
  * Neurologic or musculoskeletal disorder prohibiting exercise
  * Major neuropsychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Global Health Score | Baseline to postoperative day 90
  The primary outcome is the difference between the baseline and 90-day global health score on the European Organization for the Research and Treatment of Cancer (EORTC) QLC-C30

SECONDARY OUTCOMES:
Presence and severity of postoperative complications | Postoperatively through to day 30 and day 90
  The presence and severity of postoperative complications at 30 and 90 days will be recorded from the patient's medical records
Postoperative hospital length of stay | Length of stay will be calculated from the date of surgery until to the date of discharge from the hospital, reported in days, assessed up to 6 months postoperatively.
  The patient's postoperative length of stay will be recorded from the medical records
Changes in functional capacity from baseline | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  Patients will perform a 6-Minute Walk Test.
Changes in self-reported physical activity from baseline | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  Changes in self-reported physical activity will be measured using the Godin Leisure-time Exercise Questionnaire
Changes in health-related quality of life from baseline | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  HRQOL will be measured using the EQ-5D Health Questionnaire
Presence and severity of symptoms | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  The presence and severity of nine common symptoms in cancer patients will be examined using the Edmonton Symptom Assessment Scale (ESAS). This self-report measure examines: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, and shortness of breath.
Changes in anxiety and depression from baseline | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  Changes in anxiety and depression will be examined using the Hospital Anxiety and Depression Scale (HADS). HADS assesses anxiety and depression through self-reporting based on the frequency of symptoms over the past week. There are 2 subscales, one for anxiety and for depression, each with 7 items. Items are scored on a 4 point Likert scale (0-3), with the subscale scores being sums of each item (0-21). A higher score is indicative of higher or worse anxiety and depression.
Changes in fatigue from baseline | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  Changes in cancer-specific fatigue will be assessed using the 13-item Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F).
Interference with occupational performance and productivity | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  The degree to which the patient's health problems interfere with occupational performance and productivity will be examined using the Work Limitations Questionnaire
Changes in multidimensional social support | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  Changes in the perceived availability of multidimensional social support will be evaluated using the Medical Outcomes Study Social Support Scale (MOS-SSS SF-20). The MOS-SSS SF-20 is a 20 item questionnaire that measures physical functioning, social functioning, mental health, current health perceptions, and pain. After reverse scoring of the appropriate items according to the MOS-SSS core scoring manual, a higher value indicates better functioning, health, and more pain in the respective measures. All measure scores are transformed linearly to scales from 0-100, with 100 being the highest score possible.
Changes in attachment (closeness in relationships with others) | Baseline, immediately preoperatively, and postoperatively at 1, 3, and 6 months
  The Experiences in Close Relationships Scale (ECR M16) will be used to examine adult attachment or closeness in both romantic and non-romantic relationships. There are two domains that are measured - attachment anxiety and avoidance. Each domain includes 8 items. Items are scored on a 7 point Likert Scale (1-7). After appropriate reverse scoring, a high score indicates higher attachment anxiety or avoidance.
Health care utilization | post-operatively at 3 and 6 months
  Health care utilization will be assessed at the postoperative 3 and 6 month time points using the Health Service Utilization Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Anand Govindarajan, MD MSc, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (2):
- Canada (2):
  - Sinai Health System - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario